CLINICAL TRIAL: NCT02480348
Title: Medtronic Polymer-Free Drug-Eluting Coronary Stent System in De Novo Native Coronary Artery Lesions
Brief Title: Medtronic RevElution Trial
Acronym: RevElution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Version 5.0, 29 JUL 2019
Record Dates: First submitted 2015-06-19; First posted 2015-06-24 (Estimated); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Drug-Eluting Stents

ARMS (1):
- Polymer-free DES (Drug Eluting Stent) (Experimental)
  Interventions: Device: Polymer-free DES (Drug Eluting Stent)

INTERVENTIONS:
Device: Polymer-free DES (Drug Eluting Stent)

SUMMARY:
The purpose of this trial is to evaluate the clinical safety and efficacy of the Polymer-Free Drug-Eluting coronary stent system for the treatment of de novo lesions in native coronary arteries with a reference vessel diameter (RVD) that allows use of stents between 2.25 and 3.50 mm in diameter.

ELIGIBILITY:
Inclusion Criteria:

* Must be an acceptable candidate for percutaneous coronary intervention, stenting, & emergent coronary artery bypass graft (CABG) surgery
* Must have evidence of ischemic heart disease
* Must require treatment of either a) a single target lesion amenable to treatment with a 2.25 mm - 3.50 mm stent OR b) two target lesions located in separate target vessels, with at least one of the target lesions amenable to treatment with a 2.25 mm - 3.50 mm mm study stent
* Target lesion(s) must be de novo lesion(s) in native coronary artery(ies)

Exclusion Criteria:

* Known hypersensitivity or contraindication to aspirin, heparin and bivalirudin, thienopyridines, cobalt, nickel, platinum, iridium, chromium, molybdenum, polymer coatings (e.g. BioLinx) or a sensitivity to contrast media, which cannot be adequately pre-medicated
* History of an allergic reaction or significant sensitivity to drugs such as zotarolimus, rapamycin, tacrolimus, everolimus, or any other analogue or derivative
* History of a stroke or transient ischemic attack (TIA) within the prior 6 months
* Active peptic ulcer or upper gastrointestinal (GI) bleeding within the prior 6 months
* History of bleeding diathesis or coagulopathy or will refuse blood transfusions
* Concurrent medical condition with a life expectancy of less than 5 years
* Currently participating in an investigational drug or another device trial that has not completed the primary endpoint
* Documented left ventricular ejection fraction (LVEF) < 30% at the most recent evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2015-12-03 (Actual); Primary Completion 2017-06-16 (Actual); Study Completion 2019-10-21 (Actual)

PRIMARY OUTCOMES:
Late lumen loss (LLL, in-stent) at 9 months post-procedure as measured by quantitative coronary angiography. | 9 months

CONTACTS AND LOCATIONS:
Locations (15):
- Australia (13):
  - Eastern Heart Clinic - Prince of Wales Hospital, Sydney, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - St. Andrew's Hospital, Adelaide, South Australia
  - Royal Adelaide Hospital, Adelaide
  - Wesley Hospital / HeartCare Partners, Auchenflower
  - Flinders Medical Center, Bedford Park
  - St. Vincent's Hospital, Darlinghurst
  - Royal Brisbane & Women's Hospital, Herston
  - Monash Medical Center, Melbourne
  - Northern Hospital, Melbourne
  - Fiona Stanley Hospital, Murdoch
  - John Hunter Hospital, New Lambton
  - Royal North Shore Hospital, St Leonards
- Institute Dante Pazzanese of Cardiology, São Paulo, Brazil
- National Heart Center Singapore, Singapore, Singapore

REFERENCES:
- [Derived] Worthley SG, Abizaid A, Kirtane AJ, Simon DI, Windecker S, Brar S, Meredith IT, Shetty S, Sinhal A, Almonacid AP, Chamie D, Maehara A, Stone GW; RevElution Investigators. First-in-Human Evaluation of a Novel Polymer-Free Drug-Filled Stent: Angiographic, IVUS, OCT, and Clinical Outcomes From the RevElution Study. JACC Cardiovasc Interv. 2017 Jan 23;10(2):147-156. doi: 10.1016/j.jcin.2016.10.020. PMID 28104208